CLINICAL TRIAL: NCT02020980
Title: A Prospective, Observational Study to Assess Pain Relief After 4 Botulinum Toxin Type A (BoNT-A) Injection Cycles in Patients With Post-stroke Lower Limb Spasticity
Brief Title: RELIEF Study: Lower Limb Pain Relief After Injection Cycles in Adults Suffering From Lower Limb Spasticity Following Stroke
Acronym: RELIEF
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-92-52120-181
Record Dates: First submitted 2013-12-19; First posted 2013-12-25 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Lower Limb Spasticity
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Post-stroke lower limb spasticity patients
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — This is an observational study designed to reflect the clinical practice in real life as closely as possible.
  Botulinum Toxin Type A (BoNT-A) injection administered according to the local Summary of Product Characteristics (SmPC) and the locally agreed treatment guidelines.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The objective of this study is to demonstrate the effect of intramuscular BoNT-A injections in relieving pain, in a broad population of patients who suffer pain as the primary problem associated with spasticity. Thus, this study will help to expand the information that is available regarding the impact of BoNT-A treatment in routine clinical practice conditions.

Treatment goals can vary greatly from one patient to another and there is no unique, single outcome that reflects the treatment benefits in all the cases. Therefore, this study with special focus on the achievement of therapeutic goals, will allow the identification of each patient's specific goals regarding the improvement of the functional outcomes, the quality of life and patient well-being.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 18 years and above
* Post-stroke lower-limb spasticity
* Prior agreement with the patient to inject BoNT-A
* If previously treated with BoNT-A, (at least 3 months interval between last injection and inclusion).
* Therapeutic goals agreed jointly with the patient
* Functional Ambulation Classification (FAC) score 2-5
* Capacity to comply with the protocol
* Written informed consent

Exclusion Criteria:

* Documented positive antigenicity to botulinum toxin
* Neuromuscular disease
* Use of medications that interfere with neuromuscular transmission
* Severe muscle atrophy in any muscle to be injected
* Any other indication that might interfere with rehabilitation or the evaluation of results
* Any non-stroke spasticity diagnosis
* Pregnancy or nursing mothers
* Previous participation in any study using Goal Attainment Scale (GAS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with post-stroke lower limb spasticity in Rehabilitation and Neurology Units of hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2014-04; Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain relief on Numeric Rating Scale | Baseline visit and every 4 months up to 16 months (Visit 5).
  Pain relief evaluated by Numeric Rating Scale (NRS). The NRS score for patient self-reporting of pain ranging from 0 (no pain) to 10 (the most severe pain).

SECONDARY OUTCOMES:
Change in Pain relief on Visual Assessment Scale | Baseline visit and every 4 months up to 16 months (Visit 5).
  Pain relief evaluated by measuring changes in Visual Assessment Scale (VAS). The VAS used a 100 mm line in which values were reported, 0 (no pain) to 10 (the most severe pain).
Responder rate using goal Attainment Scale | Every 4 months up to 16 months (Visit 5).
  Responder rate assessed on the Goal Attainment Scale (GAS). GAS is a 5-point scale, with the degree of attainment captured for each goal area.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (28):
- Spain (28):
  - Hospital Marítimo Oza, A Coruña
  - Hospital General de Albacete, Albacete
  - Hospital de Basurto, Bilbao
  - Hospital de Cruces, Bilbao
  - Hospital de Galdácano, Bilbao
  - Hospital Gorliz, Bilbao
  - Hospital Guadalajara, Guadalajara
  - Hospital Dr Negrín, Las Palmas de Gran Canaria
  - Hospital Insular, Las Palmas de Gran Canaria
  - Hospital San Pedro, Logroño
  - Fundación Jimenez Díaz, Madrid
  - Hospital 12 Octubre, Madrid
  - Hospital Alcorcón, Madrid
  - Hospital General de Móstoles, Madrid
  - Hospital Principe de Asturias de Alcalá de Henares, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Ourense, Ourense
  - Hospital Son Espases, Palma de Mallorca
  - Clinica Ubarmin, Pamplona
  - Hospital Virgen de la Vega, Salamanca
  - Hospital de Donosti, San Sebastián
  - Hospital de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Canarias, Santa Cruz de Tenerife
  - Hospital Virgen de la Salud, Toledo
  - Hospital Reina Sofía, Tudela
  - Hospital Clinico Valladolid, Valladolid
  - Hospital Xeral de Vigo, Vigo
  - Hospital Universitario de Alaba, Vitoria-Gasteiz